CLINICAL TRIAL: NCT00040404
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Finding Study to Assess the Efficacy and Safety of CEP-1347 in Patients With Parkinson's Disease
Brief Title: Safety and Efficacy Study of CEP-1347 in the Treatment of Parkinson's Disease
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Unlikely to provide evidence of significant effect
Sponsor: Cephalon (Industry)
Collaborators: H. Lundbeck A/S (Industry); The Parkinson Study Group (Network)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C1347c/204/PD/US-CA
Record Dates: First submitted 2002-06-26; First posted 2002-06-27 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Idiopathic Parkinson's disease; Idiopathic Parkinson disease; Parkinson's disease, idiopathic
MeSH Terms: conditions — Parkinson Disease | interventions — 3,9-bis((ethylthio)methyl)-K-252a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CEP-1347 10mg (Experimental): CEP-1347 was administered at a dosage of 10mg twice daily (bid); capsule strengths were 5, 12.5, and 25 mg. Each patient took 2 capsules at each dosing time, approximately 12 hours apart, within 30 minutes after the morning and evening meals) for a total of 4 capsules per day.Patients were randomly assigned to CEP-1347 or placebo treatment in a 1:1:1:1 ratio. A blocked randomization scheme was used to ensure approximately equal numbers of patients in each of the 4 treatment groups at each center.
  Interventions: Drug: CEP-1347 10mg
- CEP-1347 25mg (Experimental): CEP-1347 was administered at a dosage of 25mg twice daily (bid); capsule strengths were 5, 12.5, and 25 mg. Each patient took 2 capsules at each dosing time, approximately 12 hours apart, within 30 minutes after the morning and evening meals) for a total of 4 capsules per day.Patients were randomly assigned to CEP-1347 or placebo treatment in a 1:1:1:1 ratio. A blocked randomization scheme was used to ensure approximately equal numbers of patients in each of the 4 treatment groups at each center.
  Interventions: Drug: CEP1347 25mg
- CEP-1347 50mg (Experimental): CEP-1347 was administered at a dosage of 50mg twice daily (bid); capsule strengths were 5, 12.5, and 25 mg. Each patient took 2 capsules at each dosing time, approximately 12 hours apart, within 30 minutes after the morning and evening meals) for a total of 4 capsules per day.Patients were randomly assigned to CEP-1347 or placebo treatment in a 1:1:1:1 ratio. A blocked randomization scheme was used to ensure approximately equal numbers of patients in each of the 4 treatment groups at each center.
  Interventions: Drug: CEP-1347 50mg
- Placebo (Placebo Comparator): Placebo capsules matching the CEP-1347 capsules were administered in the same manner.
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Drug: CEP-1347 10mg — CEP-1347 10mg, a K252a derivative, retains neuroprotective properties
  Arms: CEP-1347 10mg
Drug: CEP1347 25mg — CEP1347 25mg, a K252a derivative, retains neuroprotective properties
  Arms: CEP-1347 25mg
Drug: CEP-1347 50mg — CEP-1347 50mg, a K252a derivative, retains neuroprotective properties
  Arms: CEP-1347 50mg
Other: Placebo Comparator — Placebo capsules matching the CEP-1347 capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to establish safety for CEP-1347 and to determine an efficacious dose in the treatment of Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the study if all of the following criteria are met:

* Willing and able to give informed consent
* Age 30 years or older at time of diagnosis of Parkinson's disease
* Have idiopathic Parkinson's disease with at least 2 cardinal signs of disease: resting tremor, bradykinesia, or rigidity
* Modified Hoehn and Yahr stage less than or equal to 2.5
* Must have had screening procedures for cancer appropriate for the patient's age and gender, within the last 12 months; or be willing to obtain such screening before randomization
* Women: are not breastfeeding
* Women: nonchildbearing potential (ie, postmenopausal or surgically sterile) or must use a medically accepted contraceptive regimen for at least 60 days before the baseline visit, and agree to continue such use throughout the duration of the study and for 30 days after the final dose of study drug. Women must be given a pregnancy test unless they are at least 2 years postmenopausal or surgically sterile.

Exclusion Criteria:

Patients will be excluded from participating in this study if 1 or more of the following criteria are met:

* Have atypical Parkinsonism due to drugs, metabolic disorders, encephalitis, or other neurodegenerative diseases
* Have confirmed diagnosis of Parkinson's disease for more than 5 years
* Have a tremor score of 3 or more in any body part
* Have any other known medical or psychiatric condition that may compromise participation in the study
* Have a history of prior malignancy (excluding basal or squamous cell cancer of the skin) within the previous 5 years
* Have an unresolved abnormal cancer screening test result before randomization
* Have greater than trace amounts of glycosuria at screening, except for known diabetic patients
* Have estimated creatinine clearance less than 50 mL/min
* Have liver function tests (LFT) greater than 3 times the upper limit of normal (ULN)
* Have any other clinically significant ECG or laboratory finding
* Have any history of malignant melanoma
* Have history of seizures (except febrile) or posttraumatic epilepsy
* Have Mini-Mental State Exam (MMSE) score ≤ 26
* Have taken another investigational drug within 60 days before the baseline visit
* Have received prior treatment with CEP-1347
* Have received treatment with agents with potentially confounding anti-Parkinson's disease effects, with specified substrates for CYP3A4/5, or with inhibitors of CYP3A4/5
* Received treatment within 6 months before the baseline visit with agents that may induce Parkinson's disease
* Are expected, within the next 3 months, to reach a level of disability sufficient to require dopaminergic therapy
* Have BECK depression score ≥ 15
* Have known or suspected sensitivity to the investigational study drugs, including B-CIT

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Actual)
Dates: Start 2002-03; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with disability using United Parkinson's Disease Rating Scale (UPDRS) | 48 months
  Number of participants with disability sufficient to require dopaminergic therapy was assessed according to the United Parkinson's Disease Rating Scale (UPDRS) Parts I and II are historical data and are designed to rate mentation, behavior and mood; Part III is done as a motor examination at the time of a visit. The UPDRS measures patient status on a scale 0, which is normal or none, to 4, which is severe or the worst scenario.

SECONDARY OUTCOMES:
Change from Baseline to 22 months in ([123I]β-CIT) Uptake Participants | Change from Baseline to 22 months
  The effect of CEP-1347 on dopaminergic transporter density using 2β-carboxymethoxy-3β-(4-iodophenyl) tropane ([123I]β-CIT) single-photon emission computed tomography (SPECT) imaging
Safety and Tolerability as assessed by the number of participants experiencing adverse events | 48 months
  Safety was assessed by adverse events (including deaths, serious adverse events, and withdrawals due to adverse events.)

CONTACTS AND LOCATIONS:
Locations (66):
- United States (56):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of Arkansas for Medical Services, Little Rock, Arkansas
  - The Parkinson's and Movement Disorders Institute, Fountain Valley, California
  - University of California Irvine, Irvine, California
  - USC, Keck School of Pharmacy, Department of Neurology, Los Angeles, California
  - California Medical Clinic for Movement Disorders, Oxnard, California
  - Department of Neurology - UC Davis Medical Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - Stanford University Medical Center, Dept. of Neurology, Stanford, California
  - The Parkinson's Institute, Sunnyvale, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Colorado Neurological Institute/Movement Disorders Center, Englewood, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Davis Building - Neurology 8-B, Jacksonville, Florida
  - University of South Florida, Harbourside Medical Tower, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Northwestern University, Department of Neurology, Chicago, Illinois
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University of Medicine/Outpatient Clinical Research Facility, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Department of Neurology, Iowa City, Iowa
  - University of Kansas Medical Center/Dept. of Neurology, Kansas City, Kansas
  - LSUHSC in Shreveport, Shreveport, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Department of Neurology, Baltimore, Maryland
  - Center for Aging, Genetics and Neurodegeneration, Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital/Neurology, Boston, Massachusetts
  - Boston University Medical Center, Department of Neurology, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Clinical Neuroscience Center, Southfield, Michigan
  - University of Minnesota, Department of Neurology, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Creighton University/Department of Neurology, Omaha, Nebraska
  - UMDNJ Robert Wood Johnson Medical Center, New Brunswick, New Jersey
  - University of Medicine and Dentistry of New Jersey/Center for Aging, Stratford, New Jersey
  - Parkinson's Disease & Movement Disorders Center of AMC, Albany, New York
  - Movement Disorders Center/North Shore - LIJ Health System, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Beth Israel Medical Center, Department of Neurology, New York, New York
  - Columbia Presbyterian Medical Center, Neurological Institute, New York, New York
  - University of Rochester, Department of Neurology, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Medical College of Ohio, Department of Neurology, Toledo, Ohio
  - Oregon Health Sciences University/Dept. of Neurology, Portland, Oregon
  - Pennsylvania Hospital/Dept. of Neurology, Philadelphia, Pennsylvania
  - Brown University/Memorial Hospital of Rhode Island/Neurology Dept., Pawtucket, Rhode Island
  - University of Tennessee Memphis, Semmes Murphy Clinic, Memphis, Tennessee
  - Parkinson's Disease Center and Movement Disorders Clinic/Baylor College of Medicine, Houston, Texas
  - Scott and White Clinic/Texas A & M University, Temple, Texas
  - University of Virginia Health System/Adult Neurology, Charlottesville, Virginia
  - Medical College of Wisconsin, Department Neurology, Milwaukee, Wisconsin
- Canada (9):
  - University of Calgary, Calgary, Alberta
  - University of Alberta - Glenrose Rehab Hospital, Edmonton, Alberta
  - London Health Sciences Center - University Campus, London, Ontario
  - Ottawa Hospital, Civic Site, Ottawa, Ontario
  - Toronto Hospital Western Division, Toronto, Ontario
  - University of Sherbrooke, Fleurimont, Quebec
  - Centre Hospitalier De L'Universite Montreal, Montreal, Quebec
  - McGill Center for Studies in Aging, Verdun, Quebec
  - Saskatoon District Health Board - Royal University Hospital, Saskatoon, Saskatchewan
- University of Puerto Rico, Clinical Research Center, San Juan, Puerto Rico

REFERENCES:
- [Derived] Schwarzschild MA, Schwid SR, Marek K, Watts A, Lang AE, Oakes D, Shoulson I, Ascherio A; Parkinson Study Group PRECEPT Investigators; Hyson C, Gorbold E, Rudolph A, Kieburtz K, Fahn S, Gauger L, Goetz C, Seibyl J, Forrest M, Ondrasik J. Serum urate as a predictor of clinical and radiographic progression in Parkinson disease. Arch Neurol. 2008 Jun;65(6):716-23. doi: 10.1001/archneur.2008.65.6.nct70003. Epub 2008 Apr 14. PMID 18413464
- [Derived] Parkinson Study Group PRECEPT Investigators. Mixed lineage kinase inhibitor CEP-1347 fails to delay disability in early Parkinson disease. Neurology. 2007 Oct 9;69(15):1480-90. doi: 10.1212/01.wnl.0000277648.63931.c0. Epub 2007 Sep 19. PMID 17881719
- See also: The Parkinson Study Group (PSG) is a non-profit, cooperative group of Parkinson's disease experts from medical centers in the United States and Canada who are dedicated to improving treatment for persons affected by Parkinson's disease. — http://parkinson-study-group.org